CLINICAL TRIAL: NCT01185496
Title: Effectiveness and Safety Study of the DexCom™ G4 Continuous Glucose Monitoring System in Children and Adolescents With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Andrew Balo/SVP, Clinical and Regulatory Affairs, and Quality Assurance, DexCom, Inc
Other Study IDs: PTL-900220
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CGM: Blinded/Unblinded CGM wear in adjunct with SMBG meter diabetes management

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the G4 System when worn for up to 7-days by children and adolescent subjects (6 to <18 years-old) with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Device performance will be primarily evaluated in terms of the proportion of G4 System values that are within ±20% of the study meter reference value for glucose levels >80 mg/dL and ±20 mg/dL at meter glucose levels <80 mg/dL. This proportion will be compared to the proportion of such points observed in the DexCom clinical study that will be used to apply for FDA approval of the G4 System (PTL 900360) for adults.

Safety data of the G4 System will also be collected and safety will be characterized by the incidence of Adverse Device Effects, Serious Adverse Device Events, and Unanticipated Adverse Device Effects experienced by study participants.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 6 to <18 years-old;
* 2. Have been diagnosed with type 1 diabetes mellitus and are on multiple daily injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII) insulin therapy;
* 3. Willing not to inject insulin or wear an insulin pump insertion set within 3 inches from the Sensor site during Sensor wear;
* 4. Willing to use only the blood glucose meter provided to them for self-monitoring of blood glucose (SMBG) during Sensor wear, and willing to adhere to the protocol-specified fingerstick schedule during home use;
* 5. Willing to participate in three consecutive 7-day Sensor wear periods;
* 6. Willing to take a minimum of 7 fingersticks per day during home use (2 for calibration purposes, 5 for comparative purposes);
* 7. Willing to refrain from the use of acetaminophen during the Sensor insertion period and for at least 24-hours prior to Sensor insertion;
* 8. Willing not to schedule an magnetic resonance (MRI) scan, computed tomography (CT) scan, or x-ray, for the duration of the study;
* 9. Both subject and guardian are able to speak, read, and write English.

Exclusion Criteria:

* 1. Have extensive skin changes/diseases that preclude wearing the Sensor on normal skin (e.g. extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites; 2. Subjects who have a known allergy to medical-grade adhesives; 3. For participants of childbearing potential: are pregnant as demonstrated by a positive pregnancy test within 72 hours of insertion (sexually active participants of childbearing potential must use birth control during this study); 4. Have a hematocrit that is less than 30%, or greater than 55%; 5. Current participation in another investigational study protocol (if a subject has recently completed participation in another drug study, the subject must have completed that study at least 30 days prior to being enrolled in this study); 6. Have any condition that, in the opinion of the Investigator, would interfere with their participation in the trial or pose an excessive risk to study staff (e.g., known history of hepatitis B or C).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This clinical study population will consist of a minimum of 64 and up to 80 subjects with a previous diagnosis of type 1 diabetes mellitus. It is desirable to achieve an equal number of subjects enrolled into each of the following four subgroups as defined in the FDA guideline for Age Ranges of Pediatric Subgroups:
  * Female children* 6-12 years-old
  * Female adolescents** 13-17 years-old
  * Male children 6-12 years-old
  * Males adolescents 13-17 years-old
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- DexCom, Inc, San Diego, California, United States